CLINICAL TRIAL: NCT02434939
Title: Low-dose Ketamine Versus Morphine for Severe Painful Sickle Cell Crises in Children at Mulago Hospital: A Randomised Controlled Trial
Brief Title: Low-dose Ketamine vs Morphine for Vaso-occlusive Crisis in Sicklers
Acronym: KEM-VOC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013/HD07/606U
Record Dates: First submitted 2015-04-22; First posted 2015-05-06 (Estimated); Results first posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-06

CONDITIONS: Sickle Cell Crisis; Acute Pain
MeSH Terms: conditions — Vaso-Occlusive Crises; Acute Pain | interventions — Ketamine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose ketamine (Experimental): Low dose ketamine 1mg/kg given as an IV infusion via syringe pump over 10 minutes. Maximum of 2 doses to be given during study period that will last 2 hours.
  Interventions: Drug: Low dose ketamine
- Morphine (Active Comparator): Morphine 0.1mg/kg given as an IV infusion via a syringe pump over 10 minutes. Maximum of 2 doses to be given during the study period that will last 2 hours.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Low dose ketamine — Children in this arm shall receive a slow infusion of ketamine at a sub-anesthetic dose and monitored for pain, vital signs and side effects for 2 hours. Records will be taken at 5, 10, 20, 40, 60, 80, 100 and 120min.
  Other Names: Ketamine hydrochrolide 50mg/ml,Nirma Pharmaceuticals (India)
  Arms: Low dose ketamine
Drug: Morphine — Children in this arm shall receive intravenous infusion of morphine at analgesic dose and then monitored for pain, vital signs and side effects for 2 hours. Records will be taken at 5, 10, 20, 40, 60, 80, 100 and 120min.
  Other Names: Morphine sulphate 10mg/ml, Martindale Pharmaceuticals (UK)
  Arms: Morphine

SUMMARY:
This clinical trial will inform of the role of Low dose ketamine in the acute treatment of severe painful sickle cell crisis in children in a day-case sickle cell centre. The primary aim is to determine whether Low dose ketamine is non inferior to morphine in the management of acute painful sickle cell crises. The specific objectives will be to determine the maximal change in NRS pain score following administration of ketamine and to examine the safety profile of ketamine compared to morphine in this population.

The investigators hypothesize that low dose ketamine will result in similar effective pain control as morphine alone and will not be associated with an increase in adverse events.

DETAILED DESCRIPTION:
Acute pain episodes associated with sickle cell disease (SCD) are very difficult to manage effectively. Opioid, phobia, tolerance, availability and side effects have been major roadblocks in our ability to provide these patients with adequate pain relief.

Ketamine is cheap, widely safe, readily available drug in low-middle income setting, with analgesic effects at sub-anesthetic doses and has a wide range of use including surgery (opioid sparing drug), burns (change of dressing ) and cancer related pain. However literature concerning its use in sickle cell crises is still limited in our setting.

This is a double-blinded, randomized control, study comparing low-dose ketamine (LDK) to morphine for acute pain control in children with sickle cell crises. A sample of 240 children will be enrolled from a population of patients with Sickle Cell Anemia aged 7-18 who present to the Mulago Referral Hospital Sickle Cell Clinic with acute painful Vaso-occlusive Crisis (VOC). To take part in the study, a patient must have a pain score of 7 and above as assessment by the treating physician in addition to the patient meeting all other study criteria.

After enrollment, the consented patient's weight in kg will be determined at the holding area with a standardized calibrated weighing scale (SECA - From National Medical Stores, Uganda) before transfer to the treatment room.

Baseline clinical parameters which include pulse rate, respiratory rate, blood pressure, temperature, oxygen saturation, level of consciousness, Numerical Rating Scale (NRS) Pain score (with 0 being no pain and 10 being the worst pain possible) and sites of VOC pain will be noted.

This will be followed by placement of a peripheral intravenous cannula, G22-G20 (this is part of standard care) with subsequent fluid load of 15mls per kg of crystalloid, repeated if required. Other non analgesic therapies will be prescribed by the primary care provider and started concurrently.

The recruited patients will then be randomized and allocated to receive Ketamine at 1mg/kg (study drug) or morphine at 0.1mg/kg (active control) through an intravenous infusion using a syringe pump(Agilia, Fresenius Kabi) over 10 minutes.

The vital signs and NRS and Ramsay sedation scores (RSS) will be reassessed and recorded at 5, 10 and 20 minutes after the end of the drug infusion. However, patient monitoring will be continuous. At 20 minutes, patients with NRS of 5 and more will be given a second dose without crossing over. Monitoring will be continued as above. If the NRS is less than 5, they will continue to be reassessed every 20 minutes (vital signs, NRS, RSS and adverse events) until either inpatient admission to the ward or up to 120 minutes after which they will be cared for by the ward team..

If they require a third dose of pain medication at any time during the study, this will be deemed as treatment failure and the treating pediatrician will be contacted to provide further pain control.

Any Ketamine (even for morphine) side effects as listed in the risks and safety section will monitored for among the study subjects and will treated by the study team.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7-18 years
* sickle cell anemia patient with severe acute painful crisis
* Parental consent and child assent where applicable

Exclusion Criteria:

* Oxygen saturations below 90% on initial assessment
* Altered conscious and mental state that hinders communication
* Current enrollment in another clinical trial involving an investigational drug.
* History of a stroke
* Hypertension,
* Increased intracranial pressure.
* Glaucoma,
* Failed/ Difficult IV access

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felix A. Lubega, MBChB, Principal Investigator — Makerere University, College of Health Sciences, Department of Anesthesia and Critical Care; Tonny S. Luggya, MMed, Study Chair — Makerere University, College of Health Sciences, Department of Anaesthesia and Critical care; Deogratias Munube, MMed, Study Director — Makerere University, College of Health Sciences, Department of Child Health and Pediatrics; Fred Bulamba, MBChB, Study Director — Makerere University, College of Health Sciences, Department of Anaesthesia and Critical care; Mithrika S De Silva, MD, Study Director — University of Sydney, Department of Peadiatrics
Locations (1):
- Sickle Cell clinic, Mulago Hospital Complex, Kampala, Uganda

REFERENCES:
- [Background] Marcus RJ, Victoria BA, Rushman SC, Thompson JP. Comparison of ketamine and morphine for analgesia after tonsillectomy in children. Br J Anaesth. 2000 Jun;84(6):739-42. doi: 10.1093/oxfordjournals.bja.a013585. PMID 10895748
- [Derived] Lubega FA, DeSilva MS, Munube D, Nkwine R, Tumukunde J, Agaba PK, Nabukenya MT, Bulamba F, Luggya TS. Low dose ketamine versus morphine for acute severe vaso occlusive pain in children: a randomized controlled trial. Scand J Pain. 2018 Jan 26;18(1):19-27. doi: 10.1515/sjpain-2017-0140. PMID 29794277

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled children with SCD aged 7-18 with severe acute VOC admitted to the Sickle cell day care center at Mulago National Refferal Hospital from June 2015 to February 2016
Pre-assignment Details: Of the 800 patients, 314 met the inclusion criteria with a further 74 excluded. these included 28 with history stroke, 17 with SPO2 < 90, 14 declined, 2 had altered mentation and 13 had undisclosed reasons. only 240 patients were randomized.
Period: Overall Study
Arm/Group | Low Dose Ketamine | Morphine
Started | 120 | 120
Completed | 83 | 71
Not Completed | 37 | 49
Not completed — Lack of Efficacy | 34 | 48
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Ketamine | Morphine | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.8 (3.4) | 11.8 (3.6) | 11.8 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 78 | 155
  Male | 43 | 42 | 85
Weight [Mean (Standard Deviation); unit: kgs] | 30.8 (11.9) | 30.0 (12.2) | 30.4 (12.1)
Medication [Number; unit: participants]
  prior medication | 31 | 42 | 73
  no prior medication | 89 | 78 | 167
Numerical Rating Scale (NRS) pain score [Mean (Standard Deviation); unit: units on a scale] — The NRS was used to measure a patient's subjective level of pain on a scale from 0 (representing no pain at all) to 10 (the worst pain imaginable)
  units on a scale | 8.9 (1.2) | 9.2 (1.0) | 9.1 (1.1)
Temperature [Mean (Standard Deviation); unit: oC] | 36.7 (0.86) | 36.8 (0.74) | 36.8 (0.8)
blood pressure [Mean (Standard Deviation); unit: mmHg]
  systolic | 113.7 (14.0) | 115.2 (15.7) | 114.4 (14.9)
  diastolic | 64.7 (12.3) | 65.2 (14.1) | 65 (13.2)
Heart rate [Mean (Standard Deviation); unit: bpm] | 95.8 (15.8) | 98.8 (17.8) | 97.3 (16.8)
SPO2 [Mean (Standard Deviation); unit: percentage of oxygen saturation] | 93.9 (4.8) | 94.7 (3.4) | 94.3 (4.1)
respiratory rate [Mean (Standard Deviation); unit: breaths/minute] | 23.8 (5.2) | 24.5 (6.4) | 24.2 (5.8)
Glasgow Coma Scale.(GCS) [Mean (Standard Deviation); unit: units on a scale] — GCS measures level of consciousness of a patient on a scale of 3(unresponsive even to deep stimulation) to 15 ( fully conscious and alert)
  units on a scale | 15 (0) | 15 (0) | 15 (0)
Hemoglobin (Hb) [Mean (Standard Deviation); unit: g/dl] | 7.6 (1.4) | 8.3 (5.3) | 8 (3.4)
site of pain [Number; unit: participants]
  Extremity | 60 | 58 | 118
  back | 18 | 27 | 45
  chest | 30 | 23 | 53
  others | 12 | 12 | 24
status [Number; unit: participants]
  discharged | 109 | 108 | 217
  Admitted | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Maximal Change in NRS Pain Scores as a Percentage of Baseline NRS Pain Score.
Description: Our primary outcome measurement was the maximum change on the verbal NRS pain scale compared with their initial score (baseline). The NRS was used to measure a patient's subjective level of pain on a scale from 0 (representing no pain at all) to 10 (the worst pain imaginable) using whole numbers. The NRS score was documented just prior to the administration of the study drug (time zero). After infusion of the study drug was complete, NRS scores were documented at 5, 10, 20, and then every 20 minutes thereafter up to 120 minutes. We stopped recording NRS scores prior to 120 minutes if the patient requested a third dose of the study drug, withdrew consent or developed a severe adverse effect.
Time Frame: 5, 10, 20,25,30, 40,45,50 60, 80, 100, 120 minutes post drug adminstration
Population: 3 patients in ketamine arm withdrew consent after 20 minutes in to the study while 1 patient in morphine arm was discontinued due to urticarial for fear of a worsened reaction if reexposed to the drug as he required a second dose
Measure: Mean (Standard Deviation); unit: percent change from baseline NRS score.
Arm/Group | Low Dose Ketamine | Morphine
Number analyzed (Participants) | 117 | 119
percent change from baseline NRS score.
  Overall | -66.4 (29.9) | -61.3 (28.7)
  Excluding Treatment failures | -81.1 (18.0) | -79.8 (16.9)
  Among Treatment failures | -33.8 (24.2) | -33.9 (19.1)
  Those still at maximal effect at 120 | -80 (18.7) | -81.7 (17.0)
Statistical Analysis 1: Comparison: Low Dose Ketamine vs Morphine; Test type: Non-Inferiority or Equivalence — a clinically significant difference in validated pain scores was defined as 1.3. assuming both treatments are on average equal, 240 patients provided 95% power to demonstrate that IV low dose ketamine is non inferior to IV morphine with a 0.05 level of significance; p = 0.18, t-test, 2 sided; Mean Difference (Final Values) = 5.5, 95% CI 2-sided [-2.2 to 13.2]

2. Secondary Outcome: Time to Maximal Analgesic Effect and Duration of Action of Ketamine
Description: Following dosage with study medication, the amount of time taken to demonstrate the maximal change in the patient's NRS pain score.
  Maximal change in NRS pain score is to be defined as the largest change from patient's baseline pain score. Duration of maximal change is how long the patient's pain score remained at this level.
Time Frame: 5, 10, 20, 40, 60, 80, 100, 120 minutes post drug administration
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Low Dose Ketamine | Morphine
Number analyzed (Participants) | 120 | 120
minutes
  time to maximal effect | 19.8 (14.4) | 34.1 (22.1)
  duration of maximal effect | 60 (28.7) | 58.5 (30.3)

3. Secondary Outcome: Incidence of Side Effects, Including Outlying Vital Signs
Description: The patient will be assessed for vital signs (blood pressure, heart rate, respiratory rate, oxygen saturation), Ramsay Sedation Scale (RSS) score at 5,10,20 minutes following medication administration and then every 20 minutes until a total of 120 minutes from the first dose of study medication. outlying vital signs recorded.( systolic Blood pressure less than 90mmHg or greater than 150mmHg, Heart rate less than 50bpm or greater than 150bpm, oxygen saturation below 90%, respiratory rate below 9breaths/minute or greater than 40breaths/minute and RSS of 1 or greater than 3) The RSS was used to asses the level of agitation or sedation caused by the intervention .the scale ranges from 1(anxious/agitated) to 6( no response to stimulus-deep sedation) with 2 being the optimal (cooperative, oriented and tranquil).A checklist for side effects like airway problems, allergic reactions, salivation, dysphoria,nystagmus, respiratory/cardiac arrest, awakening hallucinations, nausea/vomiting was used
Time Frame: 5, 10, 20, 40, 60, 80, 100, 120 minutes post drug administration
Measure: Number; unit: participants
Groups:
- Morphine: Morphine 0.1mg/kg given as an IV infusion via a syringe pump over 10 minutes . Maximum of 2 doses to be given during the study period that will last 2 hours.
  Morphine: Children in this arm shall receive intravenous infusion of morphine at analgesic dose and then monitored for pain, vital signs and side effects for 2 hours. Records will be taken at 5, 10, 20, 40, 60, 80, 100 and 120min.
Arm/Group | Low Dose Ketamine | Morphine
Number analyzed (Participants) | 120 | 120
participants | 45 | 4

4. Secondary Outcome: Incidence of Treatment Failure by Treatment Group.
Description: Requiring more than two doses of the study medication provided for adequate pain control
Time Frame: 120 minutes
Measure: Number; unit: participants
Arm/Group | Low Dose Ketamine | Morphine
Number analyzed (Participants) | 120 | 120
participants | 34 | 48
Statistical Analysis 1: Comparison: Low Dose Ketamine vs Morphine; Test type: Non-Inferiority or Equivalence — A clinically meaningful difference in validated pain scores was defined as 1.3.Assuming both treatments are on average equal, a sample size of 240 patients (120 per group) provided 95% power to demonstrate that IV LDK is non-inferior to IV morphine with a 0.05 level of significance; p = 0.07, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 5, 10, 20,25, 30, 40,45,50,60,80,100, 120 minutes post infusion
Arm/Group | Low Dose Ketamine | Morphine
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120
Other Adverse Events (participants affected / at risk) | 45/120 | 4/120
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Ketamine (N=120) | Morphine (N=120)
nystagmus (Eye disorders) | 18 (18) | 0 (0) — involuntary repetitive eye movement
dysphoria (Nervous system disorders) | 14 (14) | 0 (0) — state of unease, anxiety, restlessness or disorientation
dizziness (General disorders) | 4 (4) | 1 (1) — feeling faint, weak or unsteady
urticaric rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — round red welts on the skin that itch intensively.
pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) — unpleasant sensation that provokes desire to scratch
Nausea & Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) — nausea- sensation of being about to vomit. vomiting- expelling of gastric contents through the mouth
over salivation (Gastrointestinal disorders) | 6 (6) | 0 (0) — produce a lot of saliva in the mouth

LIMITATIONS AND CAVEATS:
single centre trial could limit generizability, ketamine specific side effects (nystagmus) led to potential unblinding and NRS and RSS not validated for use

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No